CLINICAL TRIAL: NCT02842437
Title: Effects of Dexmedetomidine on Respiratory Function and Inflammatory Responses in Patient With Sepsis Undergoing Cleaning Focus of Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XM2015071
Record Dates: First submitted 2016-07-12; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Organ Protection
Keywords: dexmedetomidine; sepsis; respiration
MeSH Terms: conditions — Sepsis; Respiratory Aspiration | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): 25 patients receive a loading infusion of dexmedetomidine (1ug/kg) for 10min follow by a maintenance infusion (0.5ug/kg·h) continued until the end of the surgery
  Interventions: Drug: dexmedetomidine
- Placebo (Placebo Comparator): 25 patients receive matching placebo （normal saline）
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: dexmedetomidine — receive a loading infusion of dexmedetomidine (1ug/kg) for 10min follow by a maintenance infusion (0.5ug/kg·h) continued until the end of the surgery
  Arms: Dexmedetomidine
Other: normal saline — receive matching placebo (equal volume of normal saline)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of dexmedetomidine on lung protection in patient with sepsis undergoing cleaning focus of infection.

DETAILED DESCRIPTION:
Sepsis is one of the most common, life-threatening medical conditions and is frequently complicated by organ failures, especially lung injury. It is well accepted that inflammatory reaction is the major cause of lung injury. Dexmedetomidine (Dex) is a novel α2-adrenoceptor agonist that is primarily used in surgical anesthesia and conscious-sedation. Recently, animal studies have shown that Dex plays an anti-inflammatory role, while it is not known whether Dex possesses any lung protective functions in patients with sepsis. Therefore, the aim of this study is to investigate the efficacy of Dex on lung protection in patient with sepsis undergoing cleaning focus of infection.

ELIGIBILITY:
Inclusion Criteria:

* The patients with sepsis requiring abdominal cleaning focus of infection
* older than 18 years
* American Society of Anesthesiologists (ASA) physical status II-IV.

Exclusion Criteria:

* Bradycardia
* Atrioventricular block
* Allergic to the drugs
* A history of respiratory disease
* Pregnancy or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The Alveolar-Arterial Oxygen Difference | Before anesthesia
  Arterial blood samples were sampled before anesthesia for the alveolar-arterial oxygen difference by using blood gas analyzer.
The Oxygenation Index | Before anesthesia
  Arterial blood samples were sampled before anesthesia for the oxygenation index by using blood gas analyzer.
The Respiratory Index | Before anesthesia
  Arterial blood samples were sampled before anesthesia for the respiratory index by using blood gas analyzer.
The Alveolar-Arterial Oxygen Difference | At 3 minutes after the skin is sutured
  Arterial blood samples were sampled at 3 minutes after the skin is sutured for the alveolar-arterial oxygen difference by using blood gas analyzer.
The Oxygenation Index | At 3 minutes after the skin is sutured
  Arterial blood samples were sampled at 3 minutes after the skin is sutured for the oxygenation index by using blood gas analyzer.
The Respiratory Index | At 3 minutes after the skin is sutured
  Arterial blood samples were sampled at 3 minutes after the skin is sutured for the respiratory index by using blood gas analyzer.

SECONDARY OUTCOMES:
Change of tumor necrosis factor-α before anesthesia and after dexmedetomidine or placebo infusion instantly | Before anesthesia and at 3 minutes after the skin is sutured
  Blood samples were sampled before anesthesia and at 3 minutes after the skin is sutured for the serum tumor necrosis factor-α，which were analyzed by using enzyme linked immunosorbent assay (ELISA).
Change of interleukin-1β before anesthesia and after dexmedetomidine or placebo infusion instantly | Before anesthesia and at 3 minutes after the skin is sutured
  Blood samples were sampled before anesthesia and at 3 minutes after the skin is sutured for the interleukin-1β，which were analyzed by using enzyme linked immunosorbent assay (ELISA).
Change of the lactic acid before anesthesia and after dexmedetomidine or placebo infusion instantly | Before anesthesia and at 3 minutes after the skin is sutured
  Arterial blood samples were sampled before anesthesia and at 3 minutes after the skin is sutured for the lactic acid by using blood gas analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yonghai, Principal Investigator — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No